CLINICAL TRIAL: NCT01416350
Title: A Single and Repeat Dose Pharmacokinetics/ Pharmacodynamics (PK/PD) Study to Characterise theBiomarker Response in Healthy Subjects Treated With the AntiinflammatoryMacrolide Azithromycin
Brief Title: A Single and Repeat Dose PK/PD Study to Characterise Biomarker Response in Healthy Subjects Treated With Azithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 115360
Record Dates: First submitted 2011-06-23; First posted 2011-08-15 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A - randomized, open-label parallel group (Active Comparator): Part A is a randomized, open-label parallel group study evaluating PK/PD of a single azithromycin dose of 250 or 1000 mg. Data from Part A will be used to assess the dose resulting in induction/inhibition of various ex vivo biomarkers relative to a 250 mg dose of azithromycin (the clinical dose used in treatment of neutrophil-induced inflammatory conditions). This information will guide the range of doses to be studied in a FTIH study of a new chemical entity.
  Interventions: Drug: Azithromycin - 250 mg; Drug: Azithromycin - 1000 mg
- Part B - repeat dose group (Active Comparator): Part B is a repeat dose study treating subjects with Azithromycin (250 mg every other day for 3 weeks), the dose approximates that used in the treatment of chronic neutrophil-related inflammatory conditions. This information will provide insight into whether the biomarker effects change over time on repeat dosing and any potential differences observed between single and repeat doses.
  Interventions: Drug: Azithromycin - 250 mg every other day for 3 weeks

INTERVENTIONS:
Drug: Azithromycin - 250 mg — Part A - A single azithromycin dose of 250 mg.
  Arms: Part A - randomized, open-label parallel group
Drug: Azithromycin - 1000 mg — Part A - A single azithromycin dose of 1000 mg.
  Arms: Part A - randomized, open-label parallel group
Drug: Azithromycin - 250 mg every other day for 3 weeks — Part B - Repeat dose study treating subjects with Azithromycin (250 mg every other day for 3 weeks), the dose approximates that used in the treatment of chronic neutrophil-related inflammatory conditions.
  Arms: Part B - repeat dose group

SUMMARY:
This is a two part protocol (Parts A and B) in healthy volunteers evaluating the pharmacokinetics/ pharmacodynamics (PK/PD) of azithromycin to investigate the usefulness of various biomarkers (e.g., Interleukin-10 (IL-10), Granulocyte macrophage colony-stimulating factor (GM-CSF), mature dendritic cell (MDC), with and without ex vivo lipopolysaccharide (LPS) stimulation) as markers of macrolide anti-inflammatory activity.

Part A is a randomized, open-label parallel group study evaluating PK/PD of a single azithromycin dose of 250 or 1000 mg. Data from Part A will be used to assess the dose resulting in induction/inhibition of various ex vivo biomarkers relative to a 250 mg dose of azithromycin (the clinical dose used in treatment of neutrophil-induced inflammatory conditions). This information will guide the range of doses to be studied in a first time in humans (FTIH) study of a new chemical entity.

Part B is a repeat dose study treating subjects with Azithromycin (250 mg every other day for 3 weeks), the dose approximates that used in the treatment of chronic neutrophil related inflammatory conditions. This information will provide insight into whether the biomarker effects change over time on repeat dosing and any potential differences observed between single and repeat doses.

DETAILED DESCRIPTION:
This is a two part protocol (Parts A and B) in healthy volunteers evaluating the pharmacokinetics/ pharmacodynamics (PK/PD) of azithromycin to investigate the usefulness of various biomarkers (e.g., IL-10, GM-CSF, MDC, with and without ex vivo lipopolysaccharide (LPS) stimulation) as markers of macrolide anti-inflammatory activity.

Part A is a randomized, open-label parallel group study evaluating PK/PD of a single azithromycin dose of 250 or 1000 mg. Data from Part A will be used to assess the dose resulting in induction/inhibition of various ex vivo biomarkers relative to a 250 mg dose of azithromycin (the clinical dose used in treatment of neutrophil-induced inflammatory conditions). This information will guide the range of doses to be studied in a FTIH study of a new chemical entity.

Part B is a repeat dose study treating subjects with Azithromycin (250 mg every other day for 3 weeks), the dose approximates that used in the treatment of chronic neutrophil related inflammatory conditions. This information will provide insight into whether the biomarker effects change over time on repeat dosing and any potential differences observed between single and repeat doses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18 and 65 years of age inclusive
* Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy
* Child-bearing potential and agrees to use one of the contraception methods
* Body weight ≥ 50 kg and body mass index (BMI) within the range 18.5 - 30 kg/m2 (inclusive)
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions
* Single QT duration corrected for heart rate by Bazett's formula (QTcB) < 450 msec.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities
* A positive pre-study drug/alcohol screen
* A positive test for HIV antibody
* History of regular alcohol consumption within 6 months of the study
* The subject has participated in a clinical trial and has received an investigational product within the 3 months
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements
* History of sensitivity to any of the study medications, or erythromycin, any macrolide or ketolide antibiotic
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period
* The subject has donated blood in the 3 months prior to the study
* Pregnant females as determined by positive serum or urine hCG test at screening or prior to dosing
* Lactating females
* Unwillingness or inability to follow the procedures outlined in the protocol
* Subject is mentally or legally incapacitated

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-03-30 (Actual); Primary Completion 2011-05-12 (Actual); Study Completion 2011-05-12 (Actual)

PRIMARY OUTCOMES:
PK/PD modelling of the time course of concentrations and inhibition/induction of relevant biomarkers including the concentration resulting in 50% induction or inhibition (IC50) | For Part A Day 1 to 15
  Parameters from PK/PD modelling of the time course of concentrations and inhibition/induction of relevant ex vivo biomarkers (e.g., MDC, GM-CSF and IL-10 with varying levels of LPS stimulation) including the IC50 along with distribution parameters (e.g., kin and kout).
Maximum inhibition/induction of relevant biomarkers and timing of this maximum | For Part A Day 1 to 15
  Maximum inhibition/induction of relevant ex vivo biomarkers (e.g., MDC, GM-CSF and IL-10) and timing of this maximum

SECONDARY OUTCOMES:
Biomarker:Clinical Dose Ratio for each relevant biomarkers | For Part B Day 1 to 35
  Biomarker:Clinical Dose Ratio (dose which would result in maximum observed concentration (Cmax) above the concentration resulting in 80% induction or inhibition (IC80) in ≥75% of patients divided by clinical dose of 250 mg) for each relevant ex vivo biomarkers.
Observed maximum inhibition/induction and its coefficient of variation (CV) | For Part B Day 1 to 35
  For each relevant biomarker, the observed maximum inhibition/induction and its coefficient of variation (CV).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- See also: Results for study 115360 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115360?search=study&study_ids=115360#rs